CLINICAL TRIAL: NCT06396507
Title: Comparing Sulfur to Different Regimes of Permethrin for the Treatment of Scabies
Brief Title: Sulfur vs. Different Regimes of Permethrin for Scabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: University of Aleppo (Other); Tishreen University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDMS-Dermatology-06-2022
Record Dates: First submitted 2023-02-15; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Scabies
Keywords: Scabies; Permethrin; Sulfur; Skin Diseases; Parasitic Diseases; Sarcoptes scabiei; scabies mite; Skin Infectious Diseases
MeSH Terms: conditions — Scabies; Skin Diseases; Parasitic Diseases; Skin Diseases, Infectious | interventions — Permethrin; Sulfur

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the five groups (Permethrin 5% P1, P2, P3, P4, and sulfur S).
  Participants will be followed every two weeks for a month to evaluate primary and secondary outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm P1 (Active Comparator): Permethrin 5% solution
  Participants randomly assigned to this group will apply the solution once, leave it on for ≥ 8 hours, rinse it, then reapply it the same way on day 8.
  Interventions: Drug: Permethrin Solution
- Arm P2 (Experimental): Permethrin 5% solution
  Participants randomly assigned to this group will apply the solution on days one, two, and three -for ≥ 8 hours each day- then rinse it (without rinsing in between these days) and reapply it on days eight, nine, and ten then rinse it.
  Interventions: Drug: Permethrin Solution
- Arm P3 (Experimental): Permethrin 5% solution
  Participants randomly assigned to this group will apply the solution on days one, two, and three -for ≥ 8 hours each day- then rinse it (without rinsing in between these days). They will reapply it on day eight and rinse it after ≥ 8 hours.
  Interventions: Drug: Permethrin Solution
- Arm P4 (Experimental): Permethrin 5% solution
  Participants assigned to this group will apply the solution on the first two days in the first week (for ≥ 8 hours each day with rinsing in between these days) and reapply it on day eight and rinse it after ≥ 8 hours.
  Interventions: Drug: Permethrin Solution
- Arm S (Experimental): Sulfur 10%+ vaseline 90 % ointment
  Participants assigned to this group will apply the ointment for three consecutive days (for ≥ 8 hours each day and without rinsing in between these days).
  Interventions: Drug: Sulfur

INTERVENTIONS:
Drug: Permethrin Solution — permethrin 5 % solution
  Other Names: Primothrin®; Permethrin®; Cidal®
  Arms: Arm P1; Arm P2; Arm P3; Arm P4
Drug: Sulfur — Sulfur 10%+ vaseline 90 % ointment
  Other Names: sulphur
  Arms: Arm S

SUMMARY:
In 2017, the World Health Organization (WHO) labeled scabies as a neglected tropical disease. It is a serious health problem especially in poor developing countries like Syria, where overcrowding, poverty, and war consequences are considered major factors for spreading the disease. Permethrin lotion or cream is the treatment of choice for scabies, and it is applied once a week for two consecutive weeks according to the global guidelines. However, most practitioners in Syria do not adhere to this standard regimen, and a variety of regimens are used instead based mostly on clinical experience. In this study, the investigators are comparing four different regimens of permethrin application and comparing Sulfur to permethrin in terms of efficacy and safety.

DETAILED DESCRIPTION:
Background:

In 2017, the World Health Organization (WHO) labeled scabies as a neglected tropical disease that affects more than 200 million people at any time. Treating scabies in developing countries constitutes a major challenge because of factors like poverty, overcrowded areas, inadequate disease education, and low adherence to proper therapy, which together can contribute to treatment failure and the spread of the disease.

These factors abundantly exist in Syria as it is considered a developing, low-income country. Moreover, the long-term Syrian war added a significant negative impact to the socio-economic status and prevalence of scabies, raising the difficulty in controlling the disease.

Several treatment options may be used for classic scabies including permethrin 5%, crotamiton 10%, sulfur (5-10%) ointment, lindane 1%, and ivermectin. There is no ideal scabicide because the treatment choice changes according to the patient's situation, and any one of the previous agents may be used alone or in combination.

Permethrin 5% lotion or cream is the treatment of choice for scabies based on a 2007 updated Cochrane review. Most of the treatment guidelines in developing countries recommend applying the drug once a week for 8-14 hours and repeating the application after seven days. According to what is published in the medical literature, this regimen of permethrin application is usually effective and sufficient without significant drug resistance yet.

Sulfur is an old preparation for scabies treatment. It is usually used as a (5-10%) precipitated ointment over the whole body for two or three consecutive nights.

Unlike most scabicides, sulfur is effective in killing both the mites and the eggs. However, it is malodorous, cloth-spotting, and can cause irritant dermatitis. Despite the little clear scientific evidence on the clinical efficacy of sulfur and the low adherence to this treatment because of its unpleasant application effects, it is still used when the patient cannot tolerate other agents. Moreover, it is considered a safe choice in treating pregnant women and children, and it can be the only feasible scabicide in poor resources communities.

Although the evidence on repeated treatment (i.e., timing and frequency) is lacking, the majority of Syrian dermatology practitioners do not follow the classical regimen in prescribing permethrin with no specific and clear fact-based explanation of this variation. Based on a nationwide survey study the investigators conducted, 66% (105/159) of the Syrian dermatology practitioners tend to use more aggressive regimens in prescribing permethrin instead of the classic one-per-week recommended regimen.

The objective of the study:

To compare the efficacy of different regimens of permethrin application (i.e., varying in timing and frequency) to sulfur as a low-cost alternative. A secondary aim is to evaluate the adverse events and adherence.

Methods:

Participants and interventions It is a prospective, multi-center, randomized controlled trial that will be conducted at the dermatology departments of three academic hospitals run by the ministry of higher education in Syria; These hospitals are located in Damascus, Aleppo, and Latakia.

Diagnosis of scabies will be established based on the criteria of the International Alliance for the Control of Scabies (IACS 2020), which has three levels of certainty for diagnosing scabies; confirmed, clinical, and suspected scabies (Appendix A). Patients who fulfill the clinical or confirmed scabies items will be recruited. The investigators will examine the patient's skin looking for burrows, small papules, and vesicles which are the primary lesions of scabies, or the secondary lesions resulting from scratching and rubbing.

The severity of pruritus will be determined using the Verbal Rating Scale from zero (no itch) to four (very severe itch) (Appendix B). On the other hand, the severity of scabies will be measured by counting the number of lesions and grading the results as follows: score 0= Free of lesions (no scabies), score 1= 10 or fewer lesions (mild), score 2= 11- 49 lesions (moderate), score 3= 50 or more lesions (severe) (Appendix C).

Interventions:

All the participants will apply the medication in the same manner; the differences will be in the frequency of applications and showers between them. Directions of use for permethrin solution and sulfur ointment will be orally explained by the investigators to all participants with the help of figures specially designed for our study. The application of the solution will be to the whole body below the neck, including soles, between fingers and toe creases, in the folds of wrist and waistline, armpits, preauricular area, on the genitals, and beneath fingernails and toenails. Nails will be cut short, and sex will be avoided during treatment. If the patient is a child, hands and feet should be rubbed well. No supplementary treatment other than the prescribed anti-scapetic treatment is allowed during the study. Hygiene instructions are advised to be strictly followed to avoid recurrence and failure of treatment. Treatment was also instructed to all family members at the same time, including washing clothes and bedsheets at 60-celsius degrees. Clothes that cannot be washed will be put in a black plastic bag for 3 days, and vacuum cleaning will be instructed for house furniture.

The five arms of the study represent four different regimens of permethrin 5% solution application and a sulfur ointment group. The first arm (P1) will serve as the control group (i.e., active comparator), which is the standard regimen of permethrin application according to global guidelines (7). Patients on this arm will apply the 5% permethrin solution on day one, rinse it after eight hours and reapply it on day eight. Patients in group two (Arm P2) will apply the same solution on days one, two, and three then rinse it (without rinsing in between these days) and reapply it on days eight, nine, and ten then rinse it similarly to the first round. Participants in group three (Arm P3) will apply the solution on days one, two, and three then rinse it (without rinsing in between these days) and reapply it on day eight then rinse it. Participants in group four (Arm P4) will apply the solution on day one then rinse it, and on day two then rinse it. Later on day eight, they will re-apply the solution again and rinse it. Participants in group five (Arm S) will apply the ointment for three consecutive days without rinsing in between these days. Each application of the solution or the ointment is left for at least 8 hours (see figure 1 in Appendix D). Enough amounts of the previous antiscabetic medications will be distributed for free to all participants to ensure adherence and adequate and proper use of medication.

Participants who have a secondary infection will be treated with azithromycin capsules 500 mg for three consecutive days.

Participant timeline:

Participants will be assessed biweekly for at least 4 weeks starting with the day of the first application of the treatment. Participants who recovered at the "first visit" two weeks after applying the treatment will be re-evaluated at the "second visit" during the fourth week to check for recurrence. Participants who did not recover at the first visit will reapply the treatment of permethrin (according to their group regimen) as for the permethrin groups or reapply the sulfur (Arm S) as for the sulfur group. Then they will be re-evaluated at the "second visit" (week 4) and again at an additional "third visit" during week 6.

Patients who do not respond to the repeated treatment or experience recurrence (i.e., the reappearance of new lesions after complete recovery) will be treated with benzyl benzoate lotion as an alternative treatment (see figure 2 in Appendix D)

Assignment of interventions Participants will be randomly assigned to the five arms of the study using a web-based random number generator (randomlists.com). Investigators in each center will allocate the participants to the proper group and give the instructions and medications to them.

No blinding will be applied due to the different regimens of applying the medication in the permethrin groups and the different pharmaceutical properties of permethrin and sulfur.

Data collection, management, and analysis

Data collection methods:

After confirming the diagnosis according to the diagnosis criteria, data will be collected by the investigators directly from the participants, In addition to the demographic data, the structured questionnaire includes the history of the complaint, presence of secondary infection, number of family members, and the severity of itching. The follow-up questionnaire is more concise and it assesses treatment outcomes and the compliance of patients and their contacts to the instructions, in addition to the assessment of the medication side effects.

Collected data will be written on a paper form then entered into an electronic form, which will be reviewed and double-checked by the principal investigator. Photos will be taken using a mobile camera before treatment and on each visit to allow visual comparison.

Statistical methods:

Counts and percentages will be used for nominal variables. Medians and interquartile ranges will represent the continuous variables. Chi-square test will be used to study the association between categorical variables and Kruskal Wallis for continuous data. The analysis will be done using SPSS 25 software primarily, along with figures illustrated using Microsoft EXCEL.

APPENDIX A: International Alliance for the Control of Scabies (IACS 2020) A.confirmed scabies

At least one of:

A1: Mites, eggs, or faeces on light microscopy of skin samples A2: Mites, eggs, or faeces visualized on an individual using a high-powered imaging device A3: Mite visualized on an individual using dermoscopy

B. Clinical scabies

At least one of:

B1: Scabies burrows B2: Typical lesions affecting male genitalia B3: Typical lesions in a typical distribution and two history features H1: Itch H2: Positive contact history

C. Suspected scabies

One of:

C1: Typical lesions in a typical distribution and one history feature C2: Atypical lesions or atypical distribution and two history features History features

APPENDIX B: Verbal rating scale of pruritus 0 = No itch

1. = Mild itching
2. = Moderate itching
3. = Severe itching
4. = Very severe itching

APPENDIX C: Rating the lesions count Score 0 = no scabies Score 1 = lesions are 10 or less /mild/ Score 2 = lesions are between 11 - 49 /moderate/ Score 3 = lesions are 50 or more /severe/

ELIGIBILITY:
Inclusion Criteria:

* Scabies participants who meet "The 2020 International Alliance for the Control of Scabies (IACS) Consensus Criteria" level A or B.
* Participants can apply the treatment themselves or by their guardians if they are children.
* Participants willing to commit to the study's requirements

Exclusion Criteria:

* Participants are younger than two years.
* Participants with other skin diseases that could interfere with their assessment.
* Participants who received treatment for scabies in the preceding month.
* Receiving treatment with corticosteroids in the preceding week.
* Pregnancy, planning for pregnancy during the study, or breastfeeding.
* Systemic infection or receiving systemic therapy for an infectious disease
* Immunocompromised Participants.
* Participants with crusted/Norwegian scabies.
* Having sensitivity or allergy to permethrin or sulfur.
* Participants with abnormal liver and kidney functions, thyroid disease, cardiac disorders, psychiatric illnesses.
* Participation of a family member, or another member of the household in the current study.
* The number of participants' households is seven or more.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Clinical Recovery | At day 14 and 28 following the intervention.
  Clinical recovery is defined as:
  * Absence of new scabietic skin lesions, AND
  * All remaining scabietic lesions are in healing, AND
  * Improvement of itch, defined by a decrease in itching grading score up to grade 0, 1, or 2 or a decrease for one grade, as for the participants who were diagnosed as grade 2 or less from the first visit.
  The variable is binary: Yes or No.

SECONDARY OUTCOMES:
Rate of adverse events | At day 14 and 28 following the intervention.
  * Stinging (Stinging sensation after the application of the drug)
  * Erythema (any erythematous lesion that appears after the application of the drug)
  * Rash (any localized or general rash that appears after the application of the drug)
  * Itching (exaggerating of itch after the application of the drug)
  * Any other unexpected adverse events
Verbal rating scale of pruritus | At day 14 and 28 following the intervention.
  0 = No itch, 1= Mild itching, 2= Moderate itching, 3= Severe itching, 4= Very severe itching.

CONTACTS AND LOCATIONS:
Locations (3):
- Syria (3):
  - University of Aleppo, Aleppo
  - Faculty of Medicine, University of Damascus, Damascus
  - University of Tishreen, Latakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walton SF, Currie BJ. Problems in diagnosing scabies, a global disease in human and animal populations. Clin Microbiol Rev. 2007 Apr;20(2):268-79. doi: 10.1128/CMR.00042-06. PMID 17428886
- [Background] Hay RJ, Steer AC, Engelman D, Walton S. Scabies in the developing world--its prevalence, complications, and management. Clin Microbiol Infect. 2012 Apr;18(4):313-23. doi: 10.1111/j.1469-0691.2012.03798.x. PMID 22429456
- [Background] Fuller LC. Epidemiology of scabies. Curr Opin Infect Dis. 2013 Apr;26(2):123-6. doi: 10.1097/QCO.0b013e32835eb851. PMID 23411418
- [Background] Strong M, Johnstone P. Interventions for treating scabies. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000320. doi: 10.1002/14651858.CD000320.pub2. PMID 17636630
- [Background] Khalil S, Abbas O, Kibbi AG, Kurban M. Scabies in the age of increasing drug resistance. PLoS Negl Trop Dis. 2017 Nov 30;11(11):e0005920. doi: 10.1371/journal.pntd.0005920. eCollection 2017 Nov. PMID 29190303
- [Background] Karthikeyan K. Treatment of scabies: newer perspectives. Postgrad Med J. 2005 Jan;81(951):7-11. doi: 10.1136/pgmj.2003.018390. PMID 15640423
- [Background] Avila-Romay A, Alvarez-Franco M, Ruiz-Maldonado R. Therapeutic efficacy, secondary effects, and patient acceptability of 10% sulfur in either pork fat or cold cream for the treatment of scabies. Pediatr Dermatol. 1991 Mar;8(1):64-6. doi: 10.1111/j.1525-1470.1991.tb00844.x. PMID 1862029
- [Background] Chosidow O. Scabies and pediculosis. Lancet. 2000 Mar 4;355(9206):819-26. doi: 10.1016/s0140-6736(99)09458-1. PMID 10711939
- [Background] Rosumeck S, Nast A, Dressler C. Ivermectin and permethrin for treating scabies. Cochrane Database Syst Rev. 2018 Apr 2;4(4):CD012994. doi: 10.1002/14651858.CD012994. PMID 29608022
- [Background] Engelman D, Yoshizumi J, Hay RJ, Osti M, Micali G, Norton S, Walton S, Boralevi F, Bernigaud C, Bowen AC, Chang AY, Chosidow O, Estrada-Chavez G, Feldmeier H, Ishii N, Lacarrubba F, Mahe A, Maurer T, Mahdi MMA, Murdoch ME, Pariser D, Nair PA, Rehmus W, Romani L, Tilakaratne D, Tuicakau M, Walker SL, Wanat KA, Whitfeld MJ, Yotsu RR, Steer AC, Fuller LC. The 2020 International Alliance for the Control of Scabies Consensus Criteria for the Diagnosis of Scabies. Br J Dermatol. 2020 Nov;183(5):808-820. doi: 10.1111/bjd.18943. Epub 2020 Mar 29. PMID 32034956
- [Background] Sharma R, Singal A. Topical permethrin and oral ivermectin in the management of scabies: a prospective, randomized, double blind, controlled study. Indian J Dermatol Venereol Leprol. 2011 Sep-Oct;77(5):581-6. doi: 10.4103/0378-6323.84063. PMID 21860157
- See also: Randomisation — http://www.randomizer.org/
- See also: Scabies Treatment & Management: Approach Considerations, Pharmacologic Therapy, Prevention — https://emedicine.medscape.com/article/1109204-treatment
- See also: Society guideline links: Scabies — https://www.uptodate.com/contents/society-guideline-links-scabies?topicRef=114369&source=see_link